CLINICAL TRIAL: NCT01243918
Title: Evaluation of Oxygen Therapy Delivery Systems in Hypoxemic Acute Respiratory Failure
Acronym: OPTI O2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty of recruitment
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10/6-D
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Acute Respiratory Failure
Keywords: Acute respiratory failure; Oxygen therapy delivery systems; Non invasive ventilation; High concentration mask; Hypoxemic pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- VNI/Optiflow, Immunodeficient patients (Experimental): VNI = non invasive ventilation
  Interventions: Other: Oxygen therapy delivery systems
- Optiflow/VNI, Immunodeficient patients (Experimental): VNI = non invasive ventilation
  Interventions: Other: Oxygen therapy delivery systems
- Ospal/Optiflow, Immunocompetent patients (Experimental)
  Interventions: Other: Oxygen therapy delivery systems
- Optiflow/Ospal, Immunocompetent patients (Experimental)
  Interventions: Other: Oxygen therapy delivery systems

INTERVENTIONS:
Other: Oxygen therapy delivery systems — T-60 (minutes) : clinical examination, blood gas, electrocardiogram; T0 / First oxygen therapy delivery system: clinical examination, blood gas, electrocardiogram, measurement of positive and expiratory pressure and FiO2; T10 : blood gas; Between T0 and T60 (every 10 minutes): clinical examination, measurement of positive and expiratory pressure and FiO2; T60 / Second oxygen therapy delivery system: clinical examination, blood gas, electrocardiogram, measurement of positive and expiratory pressure and FiO2; T70 : blood gas; Between T60 and T120 (every 10 minutes): clinical examination, measurement of positive and expiratory pressure and FiO2; T120: clinical examination, blood gas, electrocardiogram, measurement of positive and expiratory pressure and FiO2

SUMMARY:
The main objective of this study is to evaluate the efficiency of the oxygen therapy delivery system Optiflow® compared to 2 others standard oxygen therapy delivery systems (Ospal®, non invasive ventilation).12 immunocompetent patients will compare the successive use of oxygen therapy delivery systems Optiflow®/Ospal® and 12 immunodeficient patients will compare the successive use of systems Optiflow®/Non invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in the intensive care unit of Nantes University Hospital
* Signed informed consent
* Patient with not hypercapnic acute hypoxemic respiratory failure
* Immunocompetent and immunodeficient patient

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Contra-indication to non invasive ventilation
* Allergy to xylocaine
* Coagulation troubles
* Tracheotomized patient
* Urgent indication to intubation
* Hypercapnic acute respiratory failure
* Acute pulmonary edema
* Face or nose malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Calcul of the ratio PaO2/FiO2 | one hour after each system used
  The main objective of this study is to evaluate the efficiency of the oxygen therapy delivery system Optiflow® compared to 2 others standard oxygen therapy delivery systems (Ospal®, non invasive ventilation) by calculating the ratio PaO2/FiO2

SECONDARY OUTCOMES:
number of participants with adverse events
  The secondary outcomes are to understand the mechanisms of action of Optiflow system and to evaluate the tolerance of this system:
  * number of adverse events: respiratory events, trophic troubles, subjective events (comfort, dryness of mucous membranes, gastric distension, preferred system), serious hemodynamic and cardiovascular events
  * impact on work of breathing: measure of respiratory frequency and blood gas
  * measure of positive and expiratory pressure
measure of respiratory frequency and blood gas
  The secondary outcomes are to understand the mechanisms of action of Optiflow system and to evaluate the tolerance of this system:
  * number of adverse events: respiratory events, trophic troubles, subjective events (comfort, dryness of mucous membranes, gastric distension, preferred system), serious hemodynamic and cardiovascular events
  * impact on work of breathing: measure of respiratory frequency and blood gas
  * measure of positive and expiratory pressure
measure of positive and expiratory pressure
  The secondary outcomes are to understand the mechanisms of action of Optiflow system and to evaluate the tolerance of this system:
  * number of adverse events: respiratory events, trophic troubles, subjective events (comfort, dryness of mucous membranes, gastric distension, preferred system), serious hemodynamic and cardiovascular events
  * impact on work of breathing: measure of respiratory frequency and blood gas
  * measure of positive and expiratory pressure

CONTACTS AND LOCATIONS:
Overall Officials: Noëlle BRULE, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France